CLINICAL TRIAL: NCT03576820
Title: Intranasal Lidocaine to Treat Pediatric Migraine in the Emergency Department
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-9278
Record Dates: First submitted 2018-06-08; First posted 2018-07-03 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Migraine
Keywords: pediatrics; intranasal lidocaine; migraine; headache; emergency department; pain
MeSH Terms: conditions — Migraine Disorders; Headache; Emergencies; Pain | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The medication and placebo doses will be prepared in the pharmacy at the study site and provided to the investigators in deidentified syringes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine (Experimental): Subjects will receive a one time dose of 20mg of 2% lidocaine (1 mL) via nasal mucosal atomizer
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Subjects will receive a one time dose of 1 mL of 0.9% sodium chloride solution via nasal mucosal atomizer.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — Baseline pain score and associated migraine symptoms (such as nausea, vomiting, photophobia, and phonophobia) will be recorded for each subject. Subjects will then receive intranasal lidocaine via atomizer. Pain scores will be reassessed at 5, 10, and 20 minutes. Improvement in associated symptoms will be reassessed at 20 minutes.
  Other Names: 2% Lidocaine Hydrochloride Solution (20 mg/mL)
  Arms: Lidocaine
Drug: Placebo — Baseline pain score and associated migraine symptoms (such as nausea, vomiting, photophobia, and phonophobia) will be recorded for each subject. Subjects will then receive 0.9% sodium chloride solution via atomizer. Pain scores will be reassessed at 5, 10, and 20 minutes. Improvement in associated symptoms will be reassessed at 20 minutes.
  Other Names: 0.9% sodium chloride solution
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the effect of intranasal lidocaine on pain score in pediatric patients with migraine. Patients with significant pain after oral analgesics and plan for intravenous (IV) abortive therapy will be asked to participate. Half of patients will be given intranasal lidocaine and the other half will be given placebo. Pain scores and associated migraine symptoms (i.e. nausea, vomiting, photophobia, phonophobia, avoidance of activities, and aura) will be monitored and compared between the groups.

DETAILED DESCRIPTION:
This will be a double-blinded, randomized-controlled trial using intranasal lidocaine to provide fast-acting pain relief in pediatric patients presenting with migraine to an urban pediatric emergency department (ED). Typically, abortive therapy for migraine in many emergency departments begins with oral analgesics such as ibuprofen and acetaminophen. However, many patients with inadequate pain relief after oral analgesics will require intravenous (IV) medications to abort their migraine symptoms. These medications can take up to thirty minutes or more for the onset of action to begin, potentially leaving patients in significant pain during that time. Also, obtaining IV access in children can be time-consuming and technically difficult, further delaying time to pain relief. Subjects will be given either intranasal lidocaine or placebo while awaiting IV placement and IV metoclopramide administration. Pain scales and associated migraine symptoms will be compared between the two arms before study medication administration and again at 5, 10, and 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be receiving IV metoclopramide because their migraine is refractory to oral analgesics, as determined by the treating physician.
* Moderate to severe headache with NRS score greater than or equal to 6
* Headache lasting between 2-72 hours
* Two of the following:

  1. non-occipital location of headache (frontal, frontotemporal, or unilateral)
  2. pulsating or throbbing quality
  3. aggravated by or causing avoidance of routine physical activity
  4. nausea, vomiting, or both
  5. photophobia and/or phonophobia (may be inferred from behavior)

Exclusion Criteria:

* unstable vital signs
* pregnancy
* lactating
* altered mental status
* developmental delay
* intractable vomiting
* first-time headache
* history of cardiac arrythmia
* previous adverse reaction or allergy to lidocaine
* non-English speaking

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Score | The NRS will be administered prior to study medication administration at baseline. As well as at 5 minutes, 10 minutes, and 20 minutes after study drug administration.
  The numeric rating scale (NRS) will be used to assess subjects' pain severity. This pain scale is numbered by increments of one, with a minimum score of zero and a maximum score of ten. With zero, as "no pain", and ten as "worst possible pain". We will compare the change of median pain score from baseline to three discrete time points after study medication administration for the patients who receive intranasal lidocaine compared to placebo. For this study, we will assume a decrease in pain score of 3 or more from baseline to any of the post study medication administration time points to be clinically significant.

SECONDARY OUTCOMES:
The Number of Subjects with Improvement of Associated Symptoms | Prior to study drug administration at baseline and 20 minutes after study drug administration.
  The presence or absence of nausea, vomiting, photophobia, phonophobia, aura, and avoidance of daily activities will be asked to each subject at baseline. At 20 minutes each subject will be asked to respond "yes" or "no" if each associated symptom has subjectively improved.
The Number of Subjects Who Receive IV Pain Medications | 1 hour
  All subjects will be ordered to receive IV metoclopramide. If a subject's pain significantly improved after intranasal drug administration and before IV metoclopramide administration, then metoclopramide will be held, as per discretion of the treating physician. At the end of the study the treating physician will document on the data collection sheet if the subject received IV pain medications.
The Number of Subjects with Rebound headache | 1 hour.
  Each subject will be asked to respond "yes" or "no" if their headache returned at 1 hour post study drug administration.
The Number of Subjects with Rebound headache after discharge | 1 week
  Each subject will be called within 1 week of discharge and asked to respond "yes" or "no" if they had rebound headache.
The Number of Patients that Would Use Their Intranasal Medication the Next Time They Have a Migraine | 1 hour
  At the end of the study all subjects will be asked if they would use their intranasal medication the next time they have a migraine

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Chou, MD, Principal Investigator — New York City Health and Hospitals Corporation
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barzegari H, Motamed H, Ziapour B, Hajimohammadi M, Kadkhodazadeh M. Intranasal Lidocaine for Primary Headache Management in Emergency Department; a Clinical Trial. Emerg (Tehran). 2017;5(1):e79. Epub 2017 Sep 16. PMID 29201961
- [Background] Smith D, Cheek H, Denson B, Pruitt CM. Lidocaine Pretreatment Reduces the Discomfort of Intranasal Midazolam Administration: A Randomized, Double-blind, Placebo-controlled Trial. Acad Emerg Med. 2017 Feb;24(2):161-167. doi: 10.1111/acem.13115. Epub 2017 Jan 30. PMID 27739142
- [Background] Yaeger J. Adding intranasal lidocaine to midazolam may benefit children undergoing procedural sedation. J Pediatr. 2011 Jul;159(1):166. doi: 10.1016/j.jpeds.2011.05.010. No abstract available. PMID 21669320
- [Background] Chiaretti A, Barone G, Rigante D, Ruggiero A, Pierri F, Barbi E, Barone G, Riccardi R. Intranasal lidocaine and midazolam for procedural sedation in children. Arch Dis Child. 2011 Feb;96(2):160-3. doi: 10.1136/adc.2010.188433. Epub 2010 Oct 27. PMID 21030365
- [Background] Maizels M, Geiger AM. Intranasal lidocaine for migraine: a randomized trial and open-label follow-up. Headache. 1999 Sep;39(8):543-51. doi: 10.1046/j.1526-4610.1999.3908543.x. PMID 11279969
- [Background] Maizels M. Intranasal lidocaine to prevent headache following migraine aura. Headache. 1999 Jun;39(6):439-42. doi: 10.1046/j.1526-4610.1999.3906439.x. PMID 11279923
- [Background] Kabbouche M. Management of Pediatric Migraine Headache in the Emergency Room and Infusion Center. Headache. 2015 Nov-Dec;55(10):1365-70. doi: 10.1111/head.12694. Epub 2015 Oct 21. PMID 26486800
- [Background] Richer LP, Laycock K, Millar K, Fitzpatrick E, Khangura S, Bhatt M, Guimont C, Neto G, Noseworthy S, Siemens R, Gouin S, Rowe BH; Pediatric Emergency Research Canada Emergency Department Migraine Group. Treatment of children with migraine in emergency departments: national practice variation study. Pediatrics. 2010 Jul;126(1):e150-5. doi: 10.1542/peds.2009-2337. Epub 2010 Jun 7. PMID 20530076
- [Background] Patterson-Gentile C, Szperka CL. The Changing Landscape of Pediatric Migraine Therapy: A Review. JAMA Neurol. 2018 Jul 1;75(7):881-887. doi: 10.1001/jamaneurol.2018.0046. PMID 29532087
- [Background] Brousseau DC, Duffy SJ, Anderson AC, Linakis JG. Treatment of pediatric migraine headaches: a randomized, double-blind trial of prochlorperazine versus ketorolac. Ann Emerg Med. 2004 Feb;43(2):256-62. doi: 10.1016/s0196-0644(03)00716-9. PMID 14747817
- [Background] Prensky AL, Sommer D. Diagnosis and treatment of migraine in children. Neurology. 1979 Apr;29(4):506-10. doi: 10.1212/wnl.29.4.506. PMID 571549
- [Background] Kudrow L, Kudrow DB, Sandweiss JH. Rapid and sustained relief of migraine attacks with intranasal lidocaine: preliminary findings. Headache. 1995 Feb;35(2):79-82. doi: 10.1111/j.1526-4610.1995.hed3502079.x. PMID 7737865